CLINICAL TRIAL: NCT02249858
Title: Palpatory and Ultrasound Assessment of Cervical Dysfunctions and the Effect of Cervical High Velocity Low Amplitude (HVLA) Technique
Status: Completed | Type: Observational
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BHS-988
Record Dates: First submitted 2014-02-11; First posted 2014-09-26 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Cervical Dysfunction
Keywords: cervical spine; OMT; HVLA; ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Cranial Vault Protocol Group: Cranial vault protocol group will receive cranial vault hold.
  Interventions: Procedure: Cranial Vault Hold
- Experimental Group: HVLA Protocol Group: HVLA protocol group will receive cervical HVLA to the key somatic dysfunction C2-C7 segment.
  Interventions: Procedure: Cervical HVLA

INTERVENTIONS:
Procedure: Cranial Vault Hold
  Groups: Control Group: Cranial Vault Protocol Group
Procedure: Cervical HVLA
  Groups: Experimental Group: HVLA Protocol Group

SUMMARY:
Osteopathic medicine is a distinct school of medicine. Osteopathic physicians evaluate the neuromusculoskeletal system and work to achieve normal body mechanics. They use palpation to identify somatic dysfunctions. After performing osteopathic manipulative treatment (OMT), such as high velocity low amplitude (HVLA), a dysfunction is reassessed by palpatory assessment. While there are studies which show the effectiveness of OMT, a challenge remains to objectively assess a somatic dysfunction.

The purpose of this study is to investigate the content validity of the palpatory examination for the cervical spine using ultrasonography and the effects of a single cervical HVLA technique. Content validity is the extent to which a measure adequately and comprehensively measures what it claims to be measuring. The Investigators aim to objectively assess diagnosis and treatment of the cervical spine.

HVLA technique employs a rapid, therapeutic force of brief duration that travels a short distance within the anatomic range of motion of a joint, and that engages the restrictive barrier in one or more planes of motion to elicit release of restriction. It is also known as a thrust technique. The goal of the treatment is the restoration of physiological motion to the dysfunctional joint.

Proper diagnosis of a joint dysfunction is important for spinal manipulation. Little assessment has been made of the clinician's ability to reliably identify a joint with biomechanical dysfunctions. Few studies attempt to address the challenge of evidence-based clinical practice. These have found the benefit of consensus training.

In a study conducted by Shaw et al., ultrasound machine was used to assess the content validity of palpatory examination and objectively assess the effect of HVLA in the lumbar spine. The investigators aim to adapt the protocol for the cervical spine, but with the addition of a control cohort. Subjects will be subjected to the cranial vault hold, which assesses the primary respiratory mechanism in and the degree of participation of each bone in the general motion of the cranium. In the experimental group, participants will be receiving cervical HVLA to the key somatic dysfunction.

The Investigators hypothesize that an ultrasound is a reliable instrument to objectively evaluate somatic dysfunction of the cervical spine. Furthermore, the investigators hypothesize that after performing cervical HVLA, the left and right articular pillars of the key somatic dysfunction vertebrae should be symmetrical compared to baseline.

DETAILED DESCRIPTION:
The osteopathic philosophy applies to manipulative treatment as well as viewing an individual as a whole entity. The neuromusculoskeletal system is important to sustaining a healthy life. The musculoskeletal system is intimately connected with all other systems of the body through both the voluntary and involuntary nervous systems. Osteopathic physicians are trained to evaluate the neuromusculoskeletal system and work to achieve normal body mechanics through the use of manual manipulative medicine.

Osteopathic physicians use palpatory examination to identify somatic dysfunctions. The accepted definition in the Glossary of Osteopathic Terminology is: "Somatic dysfunction is an impaired or altered function of related components of the somatic (body framework) system: Skeletal, arthrodial, and myo-fascial structures, and related vascular, lymphatic and neural elements". Physicians assess for texture changes, asymmetry, restriction of motion, and tenderness. After performing OMT, such as HVLA, a dysfunction is reassessed by palpatory assessment once again. While there are studies which show the effectiveness of OMT, a challenge remains to objectively assess a somatic dysfunction.

According to the Glossary of Osteopathic Terminology, HVLA technique is defined as "An osteopathic technique employing a rapid, therapeutic force of brief duration that travels a short distance within the anatomic range of motion of a joint, and that engages the restrictive barrier in one or more planes of motion to elicit release of restriction. It is also known as a thrust technique". The goal of the treatment is the restoration of physiological motion to the dysfunctional joint. In the past, osteopathic manipulation was synonymous with the thrust technique. This may have been because this technique can be taught by accurately describing the nature of the restriction and providing techniques for treating the dysfunction.

Proper diagnosis of a joint dysfunction is important for spinal manipulation. However, little assessment has been made of the clinician's ability to reliably identify a joint with biomechanical dysfunctions. Few studies attempts to address the challenge of evidence-based clinical practice. In a study by Degenhardt et al., investigators looked into the inter-observer reliability of the osteopathic palpatory tests. While the study showed that consensus training did show some improvement in the inter-observer reliability, many previously published studies failed to show a level of reproducibility that supports the use of palpation in evidence-based clinical practice. Najm et al. systematic review paper reasoned that one of the challenges behind evaluating the validity of palpatory assessment is due to the lack of a reference standard measuring means. The reference standard can be used to measure the findings made by palpation.

In a study conducted by Shaw et al. they were able to use an ultrasound machine to assess the content validity of palpatory examination as well as to provide objective evidence of the effect of HVLA on somatic dysfunction in the lumbar spine. We aim to adapt their protocol for the cervical spine. The study conducted by Shaw et al. did not have a control group. In our study, we aim to have a control group which will not be getting treatment in the cervical spine. The control group will be subjected to the cranial vault hold which is generally used to assess the primary respiratory mechanism in the cranium and degree of participation of each bone in the general motion of the cranium. In the experimental group, participants will be receiving cervical HVLA to the key somatic dysfunction segment. Based on Shaw et al. study, we hypothesize that an ultrasound is a reliable instrument to objectively evaluate somatic dysfunction of the cervical spine. Furthermore, we hypothesize that after performing cervical HVLA, the left and right articular pillars of the key somatic dysfunction vertebrae should be symmetrical compared to baseline.

Previous studies show certain effects observed after an HVLA manipulation. In a systematic review paper by Hegedus et al., it was found that after a single spinal joint mobilization, there were temporary neurophysiological effects for approximately 5 minutes or less. Studies that have revealed the neurophysiological effects of spinal manual therapy have caused a paradigm shift away from a strict biomechanical model. This is important because the neurophysiological effects include pain-related measures, changes in skin conductance, changes in skin temperature and improvements in range of motion with neural tensioning. In a study performed by Martinez-Segura et al., it was found that a single cervical HVLA manipulation was more effective in reducing neck pain at rest and increasing active cervical range of motion than a control mobilization procedure in subjects suffering from mechanical neck pain.

This research design holds significant importance. It can potentially prove intra- and inter-examiner reliability of palpatory assessment. In addition, ultrasonography can be used as a reference standard for evaluating somatic dysfunctions. Furthermore, this study will enable investigators to quantify the palpatory assessment and the extent to which HVLA has an effect on a key somatic dysfunction in the cervical spine. Using an ultrasound machine for the study holds many advantages. It is relatively safe and noninvasive. It enables investigators to visualize the cervical anatomy without any radiation and minimal harm to the participants. Using a cervical goniometric device, investigators will observe how the osteopathic techniques that are utilized in this study will affect active range of motion. The total time of participation is 60 minutes, and the change in range of motion from baseline to 1 hour following the intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic and healthy participants with not contraindications to HVLA
* no local metastases
* no osseous or ligamentous disruption
* no apprehension on the part of the participant

Exclusion Criteria:

* contraindications to HVLA
* diagnosis of fibromyalgia syndrome
* neck or back or cervical spine pain
* herniated nucleus pulposus
* bone diseases (such as osteoporosis)
* rheumatoid arthritis
* Down Syndrome
* prior surgery on back
* any cervical radiculopathy
* if rotation of the head and neck causes dizziness, lightheadedness or pain
* dislocation of the dens associated with rupture or laxity of the transverse ligament of the atlas.
* advance carotid disease
* recent history of seizures
* stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be 1st and 2nd year NYIT-COM medical students. 52 students will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion | Change in baseline in cervical range of motion
  Measured rotation of the cervical spine

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Flaum, DO, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York, United States

REFERENCES:
- [Background] Burns DK, Wells MR. Gross range of motion in the cervical spine: the effects of osteopathic muscle energy technique in asymptomatic subjects. J Am Osteopath Assoc. 2006 Mar;106(3):137-42. PMID 16585381
- [Background] Hegedus EJ, Goode A, Butler RJ, Slaven E. The neurophysiological effects of a single session of spinal joint mobilization: does the effect last? J Man Manip Ther. 2011 Aug;19(3):143-51. doi: 10.1179/2042618611Y.0000000003. PMID 22851877
- [Background] Martinez-Segura R, Fernandez-de-las-Penas C, Ruiz-Saez M, Lopez-Jimenez C, Rodriguez-Blanco C. Immediate effects on neck pain and active range of motion after a single cervical high-velocity low-amplitude manipulation in subjects presenting with mechanical neck pain: a randomized controlled trial. J Manipulative Physiol Ther. 2006 Sep;29(7):511-7. doi: 10.1016/j.jmpt.2006.06.022. PMID 16949939
- [Background] Najm WI, Seffinger MA, Mishra SI, Dickerson VM, Adams A, Reinsch S, Murphy LS, Goodman AF. Content validity of manual spinal palpatory exams - A systematic review. BMC Complement Altern Med. 2003 May 7;3:1. doi: 10.1186/1472-6882-3-1. Epub 2003 May 7. PMID 12734016
- [Background] Potter L, McCarthy C, Oldham J. Intraexaminer reliability of identifying a dysfunctional segment in the thoracic and lumbar spine. J Manipulative Physiol Ther. 2006 Mar-Apr;29(3):203-7. doi: 10.1016/j.jmpt.2006.01.005. PMID 16584944
- [Background] Degenhardt BF, Snider KT, Snider EJ, Johnson JC. Interobserver reliability of osteopathic palpatory diagnostic tests of the lumbar spine: improvements from consensus training. J Am Osteopath Assoc. 2005 Oct;105(10):465-73. PMID 16314679
- [Background] Shaw KA, Dougherty JJ, Treffer KD, Glaros AG. Establishing the content validity of palpatory examination for the assessment of the lumbar spine using ultrasonography: a pilot study. J Am Osteopath Assoc. 2012 Dec;112(12):775-82. doi: 10.7556/jaoa.2012.112.12.775. PMID 23212428
- [Background] Wood TG, Colloca CJ, Matthews R. A pilot randomized clinical trial on the relative effect of instrumental (MFMA) versus manual (HVLA) manipulation in the treatment of cervical spine dysfunction. J Manipulative Physiol Ther. 2001 May;24(4):260-71. doi: 10.1067/mmt.2001.114365. PMID 11353937
- [Background] Gupta A, Kaur K, Sharma S, Goyal S, Arora S, Murthy RS. Clinical aspects of acute post-operative pain management & its assessment. J Adv Pharm Technol Res. 2010 Apr;1(2):97-108. PMID 22247838